CLINICAL TRIAL: NCT07388602
Title: A Phase 3 Randomized, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of SCTC21C in Combination With Bortezomib, Cyclophosphamide, and Dexamethasone Versus Bortezomib, Cyclophosphamide, and Dexamethasone in Patients With Newly Diagnosed Systemic Light-Chain Amyloidosis
Brief Title: A Study to Evaluate the Safety and Efficacy of SCTC21C in Combination With Bortezomib, Cyclophosphamide, and Dexamethasone in Patients With Newly Diagnosed Systemic Light-Chain Amyloidosis (NDSLCA)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCTC21C-B301
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Bortezomib; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTC21C + VCd (S-VCd) (Experimental)
  Interventions: Drug: SCTC21C; Drug: Bortezomib; Drug: Dexamethasone; Drug: Cyclophosphamide
- VCd (Active Comparator)
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: SCTC21C — Pharmaceutical form: Solution for infusion； Route of administration: Subcutaneous
  Arms: SCTC21C + VCd (S-VCd)
Drug: Bortezomib — Pharmaceutical form: Lyophilized powder for injection； Route of administration: Subcutaneous
Drug: Dexamethasone — Pharmaceutical form: Tablets, ampoules or vials for injection； Route of administration: Oral/Intravenous
Drug: Cyclophosphamide — Pharmaceutical form: Tablets, ampoules or vials for injection； Route of administration: Oral/Intravenous

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SCTC21C plus cyclophosphamide, bortezomib and dexamethasone (VCd) compared with VCd alone in treatment of newly diagnosed amyloid light chain (AL) amyloidosis participants.

DETAILED DESCRIPTION:
This study comprises two phases: Part 1 is the safety run in, while Part 2 is a randomized, controlled, open-label, multicenter study. Both parts are divided into three stages: the screening period (up to 28 days before first dose/randomization), the treatment period (from Cycle 1 [28 days] Day 1 and continues until disease progression or unacceptable toxicity), and the follow-up period (Postintervention). Safety endpoints include treatment-emergent adverse events , treatment-related adverse events, serious adverse events, clinical laboratory tests, vital signs, physical examinations, electrocardiograms , etc. Efficacy endpoints include Overall Complete Hematologic Response (CHR)，objective response rate (ORR), Hematologic Very Good Partial Response (VGPR) or Better Rate, Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of amyloidosis based on detection by immunohistochemistry and polarizing light microscopy of green bi-refringent material in congo red stained tissue specimens or characteristic electron microscopy appearance;
* Measurable disease of amyloid light-chain (AL) amyloidosis;
* One or more organs impacted by AL amyloidosis according to consensus guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2

Exclusion Criteria:

* Prior therapy for AL amyloidosis;
* Other amyloidosis;
* Uncontrolled infection.
* Subjects with conditions that may affect safety or efficacy assessments include, but are not limited to, cardiovascular, respiratory, endocrine/metabolic, immune system, hepatic, gastrointestinal (such as gastrointestinal bleeding, perforation, ulcers, etc.), and malignant neoplasms, and are deemed clinically significant by the investigator.
* Subjects who have undergone major surgery or experienced significant trauma within 4 weeks prior to the first use of the investigational drug, or who require elective surgery during the trial period.
* Received a live or attenuated vaccine within 30 days prior to the first dose; Female subjects who are currently breastfeeding.
* Subjects with mental disorders or poor compliance, or other circumstances deemed unsuitable for participation in this study by other investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Overall Complete Hematologic Response (CHR) | Up to approximately 50 months after the First Participant In (FPI)
  Overall CHR rate was defined as percentage of participants who achieved CHR, according to the International Amyloidosis Consensus Criteria.

SECONDARY OUTCOMES:
Major Organ Deterioration Progression-Free Survival (MOD-PFS) | Up to approximately 50 months after the FPI
  MOD-PFS was defined as duration from the date of randomization to either hematologic progression, or major organ deterioration (clinical manifestation of cardiac failure or renal failure), or death, whichever occurred first.
Percentage of Participants Who Achieved Complete Hematologic Response (CHR) at 6 Months | Month 6
  CHR rate was defined as percentage of participants who achieved CHR, according to the International Amyloidosis Consensus Criteria.
Duration of Complete Hematologic Response (CHR) | Up to approximately 50 months after the FPI
  Duration of CHR was defined as the time between the date of initial documentation of CHR to the date of first documented evidence of hematologic progressive diseased.
Hematologic Very Good Partial Response (VGPR) or Better Rate | Up to approximately 50 months after the FPI
  Hematologic VGPR or Better Rate was defined as percentage of participants who achieved hematologic Complete response (CR) or VGPR.
Overall Survival (OS) | Up to approximately 50 months after the FPI
  Overall survival (OS) was measured from the date of randomization to the date of the participant's death.
Adverse Events | Up to approximately 50 months after the FPI
  Treatment-emergent adverse events/serious adverse events

OTHER OUTCOMES:
PRO: EQ-5D-5L | Up to approximately 50 months after the FPI
  Health state utility and health status will be assessed using the European Quality of Life Group questionnaire with 5 dimensions and 5 levels per dimension (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China